CLINICAL TRIAL: NCT07385872
Title: Feasibility and Performance of a Novel Concept for Internal Fixation of a Peripheral Nerve Block Catheter in Patients Undergoing Femoral Amputation
Brief Title: Performance of a Novel Concept for Internal Fixation of a Novel Peripheral Nerve Block Catheter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Hvidovre University Hospital (Other); Nordstar Medical (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Ethical Committee nr: 16098489
Record Dates: First submitted 2026-01-15; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Primary Condition: Nerve Block; Secondary Condition: Catheter Displacement; Focus of Study: Sciatic Nerve
Keywords: Sciatic Nerve Block; Peripheral Nerve Catheter; Catheter Migration; Internal Fixation Device; Proof-of-Concept Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sciatic Nerve Catheter (Experimental): All participants will receive the prototype fixation catheter placed near the sciatic nerve distal to the planned amputation line.
  Interventions: Device: Novel Internal Fixation Nerve Block Catheter - Sciatic Nerve
- Saphenous Nerve Catheter (Experimental): If the planned amputation line is high enough on the femur to allow for distal placement, participants will also receive a second prototype fixation catheter near the saphenous nerve.
  Interventions: Device: Novel Internal Fixation Nerve Block Catheter - Saphenous nerve

INTERVENTIONS:
Device: Novel Internal Fixation Nerve Block Catheter - Sciatic Nerve — A peripheral nerve block catheter prototype featuring internal fixation to prevent dislocation and a rapid-deployment system.
  Catheters are placed under ultrasound guidance.
  Arms: Sciatic Nerve Catheter
Device: Novel Internal Fixation Nerve Block Catheter - Saphenous nerve — Placement of the saphenous catheter is contingent upon an amputation line that allows for placement below the surgical site (distal to the cut).
  Arms: Saphenous Nerve Catheter

SUMMARY:
The goal of this study is to test a new type of nerve block catheter (a thin, flexible tube used to deliver pain medication). Researchers want to see if this new design stays in its original position better than current catheters and if it is easy for doctors to use.

The main questions the study aims to answer are:

Does the catheter tip stay in the correct position over time without moving or slipping (dislocation)?

Can the catheter be placed quickly and accurately using the new deployment system?

Researchers will test this prototype in a small group of participants. There is no comparison group for this initial study.

Participants will:

Have the catheter placed near a nerve in their leg a few days before a scheduled femoral (leg) amputation.

Undergo imaging or checks to see if the catheter has moved.

Have the catheter removed just before their scheduled surgery.

The catheter will be placed in an area of the leg that is already scheduled to be removed during surgery. This ensures that the study carries minimal risk to the participants.

DETAILED DESCRIPTION:
Background and Rationale Peripheral nerve blocks are a standard of care for regional anesthesia; however, traditional catheters are prone to secondary dislocation (slipping out of place), which leads to inadequate pain control. This study evaluates a novel prototype catheter designed with an internal fixation mechanism intended to secure the catheter tip at the target site. Additionally, the system utilizes a refined deployment mechanism designed for rapid and precise placement by the clinician.

Study Objective The primary objective of this pilot study is to evaluate the stability and migration rate of the catheter tip over a multi-day period. Secondarily, the study will assess the technical feasibility and speed of the deployment system.

Study Design and Safety Model This is a single-arm, non-randomized, proof-of-concept trial. To ensure maximum participant safety during the testing of this new hardware, the study utilizes a femoral amputation model.

The catheter will be placed in participants who are already scheduled for a femoral amputation. The insertion site and the final position of the catheter tip will be located distal to (below) the anticipated surgical amputation line. This ensures that the tissue involved in the study is part of the limb intended for removal, thereby minimizing any long-term risk of nerve injury or local tissue complications for the participant.

Procedures

Baseline & Placement: Eligible participants will have the prototype catheter placed via ultrasound guidance several days prior to their scheduled surgery. The time required for deployment will be recorded.

Monitoring Period: The position of the catheter tip will be monitored at set intervals using ultrasound imaging to track any migration or dislocation from the initial placement site.

Removal: The catheter will be removed in the operating room immediately prior to the commencement of the scheduled amputation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for elective transfemoral amputation
* Able and willing to provide informed consent

Exclusion Criteria:

* Known allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Catheter Dislocation Distance | From initial placement (Day 0) to immediately prior to amputation surgery (typically 48-72 hours).
  The absolute distance (in millimeters) between the position of the catheter delivery orifice at initial placement and its position just before removal. The position is verified by ultrasound imaging using hydrodissection with a local anesthetic bolus to identify the orifice.

SECONDARY OUTCOMES:
Time on Task | At time of procedure (Day 0)
  Time required for catheter placement, measured from initiation of skin disinfection to final skin fixation using a stopwatch (seconds).
Primary Placement Success Rate | At time of procedure (Day 0)
  Proportion of successful primary catheter placements, defined as the accurate position of the delivery orifice verified by ultrasound
Catheter Clinical Performance (Sensory Block) | Day 0 (preprocedure and postprocedure), day 1, day 2, and day 3.
  Sensitivity to a cooled vial (5°C) over the cutaneous innervation area (Tibial/Peroneal for sciatic; Saphenous for saphenous nerve).
Catheter Retraction Force | Day 3 (just before surgery)
  The force required for catheter removal, measured with a digital handheld force transducer (Newtons).
Pain Intensity (NRS) | Day 0, Day 1, Day 2 and Day 3
  Participant-reported pain at rest using a Numeric Rating Scale (0-10, where 0 is no pain and 10 the worst thinkable pain)
Cumulative Opioid Consumption | Day 0 to day 3 (Entire study duration)
  Total intravenous (IV) morphine equivalents administered while the catheter is in place.
Incidence of Adverse Events | Day 0 to day 3 (Entire study duration)
  Number and nature of complications including infection, back-leakage, or device-related issues.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer C Jørgensen, MD, PhD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Hvidovre Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Whether individual participant data will be shared has not yet been determined. The study evaluates novel design principles and mechanical fixation mechanisms for which intellectual property (IP) protection is currently being sought or finalized. A decision regarding the sharing of de-identified data will be made once the proprietary interests of the device design are fully secured and the primary feasibility analysis is complete.

REFERENCES:
- [Background] Carvalho BY, Mariano ER. Continuous vs. single-injection peripheral nerve blocks: A prospective cohort study comparing procedural time and personnel cost. Open Anesthesiol J. 2015;9:1-5.
- [Background] Martin N, Davis CJ. Evidence from masked-priming that initial identification of brand names is via abstract letter identities. Br J Psychol. 2019 Nov;110(4):745-768. doi: 10.1111/bjop.12362. Epub 2019 Jan 4. PMID 30613945
- [Background] Baillie J, Lankshear A. PATIENTS' AND RELATIVES' EXPERIENCES OF PERITONITIS WHEN USING PERITONEAL DIALYSIS. J Ren Care. 2015 Sep;41(3):177-86. doi: 10.1111/jorc.12118. Epub 2015 Feb 27. PMID 25727142
- [Background] Hauritz RW, Hannig KE, Balocco AL, Peeters G, Hadzic A, Borglum J, Bendtsen TF. Peripheral nerve catheters: A critical review of the efficacy. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):325-339. doi: 10.1016/j.bpa.2019.07.015. Epub 2019 Jul 22. PMID 31785718
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354